CLINICAL TRIAL: NCT01063621
Title: Phase 3 Study of KW-6500 (Safety Study for Extended Long-Term Self-Injection at Home in Patients With Parkinson's Disease)
Brief Title: Extended Long-Term Safety Study of KW-6500
Acronym: 6500-005
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6500-005
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

ARMS (1):
- KW-6500 (Experimental)
  Interventions: Drug: KW-6500

INTERVENTIONS:
Drug: KW-6500 — Subcutaneous injection of 1 to 6 mg for the OFF state during 52 weeks
  Other Names: Apomorphine hydroshloride (USAN)

SUMMARY:
This is a extended long-term safety study in Parkinson's disease patients who have motor response complications on levodopa therapy and completed 12 weeks administrations of KW-6500 in 6500-004 study. The safety and efficacy of long-term subcutaneous self-injections of KW-6500 are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent
* Patients who have completed the 6500-004 study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-01; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Adverse events and related adverse events | From first administration of study drug through Study Week 52

SECONDARY OUTCOMES:
Time to expression of the ON state, continuous time of the ON state, raw score change and percent score change in UPDRS part III, response ratio, and UPDRS part II score | From first administration of study drug through Study Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Tōon, Ehime, Japan